CLINICAL TRIAL: NCT01885091
Title: Kinerase® Interactive Skin-care Study: A Multicentre, Phase IV, Single-arm, Open-label Trial to Evaluate the Efficacy and Safety of Kinetin, N6-furfuryladenine, 0.1% for Treatment of Cutaneous Facial Photodamage
Brief Title: Efficacy and Safety Study of Kinerase® for Treatment of Cutaneous Facial Photodamage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini (Thailand) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K.I.S.S
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Skin Roughness; Mottling; Blotchiness; Pigmentation; Fine Wrinkles
MeSH Terms: interventions — Kinetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kinerase (Experimental)
  Interventions: Other: Kinerase

INTERVENTIONS:
Other: Kinerase

SUMMARY:
The purpose of the K.I.S.S. study is to evaluate the efficacy of Kinerase® Cream (Kinetin 0.1%) in Thai patients, on the basis of the severity and clinical signs of facial photodamage.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects older than 35 years of age and less than 65 years of age.
2. Subjects with mild, moderate or severe facial photodamage as assessed by a 10-point scale.
3. Subjects willing to sign an informed consent and adhere to all protocol requirements.

Exclusion Criteria:

1. Male and female subjects with suspected porphyria, systemic or cutaneous erythematosus lupus, or any other photosensitizing disorder or drug-induced photosensitization.
2. Subjects with chronic or recurring skin disease or disorder.
3. Subjects with any active infectious skin disorder (Herpes simplex, molluscum contagiosum, and facial warts).
4. Subjects with skin cancer of the facial tissues.
5. Subjects who have received any laser/ intense pulsed light (IPL) / chemical peel in the 2 months preceding the screening visit.
6. Subjects with a history of topical and/or oral isotretinoin use, 6 months prior to the screening visit.
7. Subjects who have been on topical Retin-A or Renova in the 2 months prior to the screening visit.
8. Subjects who have used topical alpha-hydroxy acid skin care products in the month preceding the screening visit.
9. Subjects currently on any anti-aging products and who wish to continue use of their products.
10. Subjects requiring concurrent treatment that would interfere with the study assessments.
11. Pregnant or lactating female subjects.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To assess the physician's evaluation and patient's self-evaluation at 12 weeks. | 12 weeks
To assess the physician's evaluation and patient's self-evaluation at 4 weeks. | 4 weeks
To assess the physician's evaluation and patient's self-evaluation at 8 weeks. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rungsima Wanitphakdeedecha, MD, MA, MSc, Principal Investigator — iSKY Innovative Skin & Laser Surgery Center
Locations (1):
- I-Sky Center Chidlom branch, Bangkok, Bangkok, Thailand